CLINICAL TRIAL: NCT01683253
Title: The REmission of the Impulse Control Disorder and the Changes of the Neuropsychiatric Characteristics After Switching Into Levodopa/Carbidopa in Patients With Parkinson's Disease Who Have Developed Impulse Control Disorders Due to the Dopamine Replacement Therapy
Brief Title: Remission of ICD by Switching Dopamine Agonist to Levodopa/Carbidopa
Acronym: REIN-PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKL004
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Impulse Control Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Levodopa; Carbidopa; Dopamine Agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (3):
- Levodopa/Carbidopa(200mg/50mg) (Experimental)
  Interventions: Drug: Levodopa/Carbidopa(200mg/50mg)
- Control A (dopaminergic agonist ) (Experimental): Parkinson patients treated with anti-Parkinson drug over 6 months.
  Interventions: Drug: Dopaminergic Agonists
- Control B (no drug) (No Intervention): Parkinson diseased patients not treated.

INTERVENTIONS:
Drug: Levodopa/Carbidopa(200mg/50mg)
  Arms: Levodopa/Carbidopa(200mg/50mg)
Drug: Dopaminergic Agonists — Treated for at least 6 months after diagnosis of Parkinson's Disease.
  Arms: Control A (dopaminergic agonist )

SUMMARY:
The purpose of this study is to see whether the ICDs(Impulse Control Disorder) are improved and neuropsychiatric traits related to ICD are changed or not when switching dopamine agonist to levodopa/carbidopa in patients with Parkinson's disease who have been treated with dopaminergic medications.

DETAILED DESCRIPTION:
* PRIMARY OBJECTIVE To evaluate the improvement of mMIDI(modified version of Minnesota Impulsive Disorders Interview,Korean version) score from the baseline to 12 weeks or LOCF(Last Observation Carried Forward)
* SECONDARY OBJECTIVE i) To evaluate the improvement of neuropsychiatric profiles from the baseline to 12 weeks or LOCF ii) To evaluate the improvement of UPDRS(Unified Parkinson's Disease Rating Scale)Score from the baseline to 12 weeks or LOCF

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of idiopathic PD according to United Kingdom Parkinson's Disease Brain Bank Criteria
* mMIDI ≥ 3 score with ICD
* Patients must be on an anti-parkinson treatment at least 6 months before screening.
* for this protocol, dopamine agonists should be included in his/her anti-parkinson treatment.
* 30years ≤ patients < 80years of age, male or female
* patients must give written informed consent before any assessment is performed

Exclusion Criteria:

* Requirement of treatment with serious cognitive disorder, behavioral disorder, or mental illness currently or in the future
* for the patients ≤ 65years: K-MMSE(korean version of Mini-Mental State Exam) ≤24, or for the patients ≥ 66years: K-MMSE ≤ 20, or the patients have dementia(incl. early dementia) even though K-MMSE score is more than 20
* Requirement of treatment more than 6times per day due to the severe motor fluctuation.
* Severe dyskinesia
* DBS(Deep Brain Stimulation)or any other surgical treatment
* History of melanoma or not-diagnostic skin trouble/skin lesions
* narrow angle glaucoma
* clinically serious surgical or medical condition
* malignant tumor
* use of other investigational drugs at the time of enrollment within 4weeks
* pregnant, nursing or lactating women
* women of child-bearing potential
* history of hypersensitivity or allergy to levodopa/carbidopa
* any serious disease according to the investigator's discretion

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mMIDI(modified Minnesota Impulsive Disorders Interview) | 12weeks
  To evaluate the improvement of mMIDI(Korean version) score from the baseline to 12 weeks or LOCF(Last Observation Carried Forward)

SECONDARY OUTCOMES:
Neuropsychiatric profile | 12 weeks
  To evaluate the improvement of neuropsychiatric profiles from the baseline to 12 weeks or LOCF
  * Neuropsychological assessment
  * General cognitive status: K-Minimental status exam(K-MMSE)
  * Psychiatric profile:
    * Neuropsychiatric inventory (K-NPI)
    * Beck depression inventory (BDI)
    * Barratt impulsiveness scale (BIS)
    * Beck anxiety inventory (BAI)
    * State-trait anger expression inventory (STAXI)
    * Obsessive compulsive inventory (OCI)
  * Evaluation of global change:
    * Patient global impression of improvement (PGI-I)
    * Clinical global impression of improvement (CGI-I)

CONTACTS AND LOCATIONS:
Overall Officials: Jinwhan Cho, MD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Sandoz Investigative Site, Anyang
  - Sandoz Investigative Site, Daegu
  - Sandoz Investigative Site, Pusan
  - Sandoz Investigative Site, Seongnam
  - Sandoz Investigative Site, Seoul

REFERENCES:
- [Derived] Lee JY, Jeon B, Koh SB, Yoon WT, Lee HW, Kwon OD, Kim JW, Kim JM, Ma HI, Kim HT, Baik JS, Cho J; (REIN-PD Investigators). Behavioural and trait changes in parkinsonian patients with impulse control disorder after switching from dopamine agonist to levodopa therapy: results of REIN-PD trial. J Neurol Neurosurg Psychiatry. 2019 Jan;90(1):30-37. doi: 10.1136/jnnp-2018-318942. Epub 2018 Oct 25. PMID 30361296